CLINICAL TRIAL: NCT02201329
Title: An Open Label Phase I Trial of Intravenous Volasertib in Combination With Subcutaneous Azacitidine in Japanese Patients With Higher-risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Brief Title: Volasertib in Combination With Azacitidine in Japanese Patients With Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.35
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; BI 6727

ARMS (1):
- A (Experimental): Volasertib escalating doses + azacitidine
  Interventions: Drug: Azacitidine; Drug: Volasertib

INTERVENTIONS:
Drug: Azacitidine — Azacitidine (subcutaneous)
Drug: Volasertib — Volasertib escalating doses (intravenous)

SUMMARY:
To identify the maximum tolerated dose or recommended dose for further development of volasertib in combination with azacitidine in Japanese patients with myelodysplastic syndromes or chronic myelomonocytic leukemia, and evaluate the safety and tolerability, pharmacokinetics and the preliminary efficacy of this combination.

ELIGIBILITY:
Inclusion criteria:

1. Patients of age >=20 and <=80 years
2. Patients with primary or treatment-related myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML), who are not eligible for hematopoietic stem cell transplantation based on the investigator's judgment, that meet one of the following criteria:

   * Intermediate-2 and high-risk MDS according to the International Prognostic Scoring System, in the setting of 5-30% bone marrow blasts
   * CMML with >= 10% marrow blasts without myeloproliferative disorder (white blood cell count of <13,000/ µL)
3. Patients with no prior azacitidine treatment, or with prior azacitidine treatment that meet one of the following criteria:

   * Patients failing to achieve haematological improvement, partial remission, marrow complete remission or complete remission after 3 cycles of azacitidine or progressed at any time after start of azacitidine
   * Patients achieved an initial response and subsequently develop disease progression or relapse
4. Eastern Cooperative Oncology Group performance status score 0 or 1 at screening
5. Signed written informed consent consistent with Good Clinical Practice.

Exclusion criteria:

1. Treatment with systemic therapy for MDS, including an investigational drug, within 14 days before the first dose of study treatment, except for lenalidomide within 12 weeks before the first dose of study treatment, or lack of recovery from any acute toxicities pertinent to the prior systemic therapy.
2. Prior treatment with volasertib
3. Contraindications for azacitidine treatment according to the manufacturer's product information
4. Known hypersensitivity to the trial drugs or its excipients
5. Concomitant malignancy currently requiring active therapy (except for hormonal/anti-hormonal treatment, e.g. in prostate or breast cancer)
6. QTcF prolongation >470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome).
7. Total bilirubin >1.5 x upper limit of normal (ULN) not related to Gilbert's syndrome, hemolysis, or secondary to MDS at screening
8. Aspartate amino transferase or alanine amino transferase >2.5 x ULN
9. Serum creatinine >1.5 x ULN at screening
10. Arterial oxygen pressure <60 torr or arterial oxygen saturation <92% (at room air)
11. Active hepatitis B or hepatitis C, or laboratory evidence of hepatitis with positive results of hepatitis B surface antigen and/or hepatitis C antibody.
12. Human immunodeficiency virus infection.
13. Severe illness or organ dysfunction involving the heart, lung, kidney, liver or other organ system, which in the opinion of the investigator would interfere with the evaluation of the safety of the study treatment including; infection requiring active treatment, poorly controlled ventricular/atrial tachyarrhythmia, use of heart pacer, unstable angina pectoris, history of myocardial infarction or severe congestive heart failure, clinically unstable cardiac or pulmonary disease
14. Any significant concurrent psychiatric disorder or social situation that according to the investigator's judgment would compromise patient's safety or compliance, interfere with consent, study participation, or interpretation of study results
15. All male patients and female patients of child bearing potential who are unwilling to use a medically acceptable method of contraception during the trial and at least 6 months after the end of study treatment (i.e. hormonal contraception, intrauterine device, condom with spermicide, etc.). Note: females are considered to be of child bearing potential unless they have been surgically sterilized or are post-menopausal (complete absence of menses for at least 12 months without other medical reasons).
16. Pregnant or nursing female patients
17. Known or suspected active alcohol or drug abuse

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Japan (4):
  - Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - Boehringer Ingelheim Investigational Site, Gunma, Maebashi
  - Boehringer Ingelheim Investigational Site, Nagasaki, Nagasaki
  - Boehringer Ingelheim Investigational Site, Tokyo, Sinagawa-ku

RESULTS

PARTICIPANT FLOW:
Groups:
- Volasertib 200 mg: The patients received Volasertib 200 mg administered by Intravenous Infusion (IV) over 60 minutes on Day 1 and Day 15 of 28-day and Azacitidine 75 mg/m^2 administered by subcutaneous injection on days 1-7 of 28 day treatment cycle.
Period: Overall Study
Arm/Group | Volasertib 200 mg
Started | 5
Completed | 0
Not Completed | 5
Not completed — Progressive Dis./Relapse/Clinical Prog. | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set included all patients who were dispensed study medication and were documented to have taken at least one dose of either Volasertib or Azacitidine.
Arm/Group | Volasertib 200 mg
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: This outcome measure presents number of participants with DLTs in the first cycle for the determination of MTD. DLT was defined as any of the following Adverse Events (AEs) considered to be related to the study drug (Volasertib and/or Azacitidine).
  1. Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 drug-related non-haematologic toxicity.
  2. Drug-related AEs that led to inability to deliver the full dose of the study drugs (Volasertib and/or Azacitidine) according to the assigned dose level within Cycle 1.
  3. Absence of haematological recovery (sustained CTCAE grade ≥3 thrombocytopenia <50000/mm^3 and/or neutropenia <1000/mm^3) after completing Cycle 1 and lasting at least until Day 57 (from Day 1 of Cycle 1) despite complete marrow blast clearance on Day 29 (<5% blasts in the bone marrow.
  4. Any other drug-related AEs that required treatment delay of ≥4 weeks between the Cycle 1 and Cycle 2 (i.e., Cycle 2 was not started until Day 57 of Cycle 1)).
Time Frame: Up to 57 days.
Population: MTD Set: This patient set included all patients in the treated set who were evaluable for MTD determination.
Measure: Number; unit: Participants
Arm/Group | Volasertib 200 mg
Number analyzed (Participants) | 5
Participants | 2

2. Primary Outcome: Maximum Tolerated Dose of Volasertib
Description: This outcome measure presents MTD of Volasertib in Combination with Azacitidine. The MTD was defined as the highest dose level at which Dose Limiting Toxicities (DLTs) were reported in not more than 1 in 6 evaluable patients during Cycle 1.
Time Frame: Up to 57 days.
Population: MTD Set: This patient set included all patients in the treated set who were evaluable for MTD determination.
Measure: Number; unit: mg
Arm/Group | Volasertib 200 mg
Number analyzed (Participants) | 5
mg | NA — On the basis of DLTs, the MTD of Volasertib administered intravenously on Days 1 and 15 in 28-day cycles in combination with Azacitidine was considered to be less than 200 mg.

3. Secondary Outcome: Overall Objective Response (OR): Complete Remission (CR), Partial Remission (PR), or Marrow CR (mCR)
Description: This outcome measure presents overall Objective Response (CR+PR+mCR). Response to treatment was evaluated according to the International Working Group (IWG) 2006 criteria. Best response was tabulated from all available data, with each patient being classified into one of the categories defined in CR, PR, mCR.
Time Frame: Up to 9 months.
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Volasertib 200 mg
Number analyzed (Participants) | 5
Participants
  Objective Response (OR) | 2
  Complete Remission (CR) | 0
  Partial Remission (PR) | 0
  Marrow Complete Remission (mCR) | 2

4. Secondary Outcome: Maximum Measured Concentration of the Volasertib 200 mg in Plasma (Cmax)
Description: This outcome measure presents maximum measured concentration of Volasertib 200 mg in plasma (Cmax).
Time Frame: -0.05 hours before drug administration and 0:30 (hours:minutes), 1:00, 1:30, 2:00, 3:00, 4:00, 24:30, 48:30, 96:30, 144:30 and 335:55 after drug administration.
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Volasertib 200 mg
Number analyzed (Participants) | 5
ng/mL | 713 (44.4)

5. Secondary Outcome: Area Under the Concentration-Time Curve of Volasertib 200 mg in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: This outcome measure presents area under the concentration-time curve of Volasertib 200 mg + Azacitidine 75 mg/m^2 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: as for outcome 4
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib 200 mg
Number analyzed (Participants) | 5
ng*h/mL | 4190 (25.4)

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last trial drug administration in the last treatment cycle or the decision of study treatment discontinuation, whichever is later, and was up to 389 days.
Arm/Group | Volasertib 200 mg
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 200 mg (N=5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 200 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Eyelids pruritus (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tongue coated (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Injection site reaction (General disorders) | 5
Oedema peripheral (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Iron overload (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.